CLINICAL TRIAL: NCT05808465
Title: Comparative Study Between Phase Contrast,Modified Simpson Rule and Myocardial Strain Analysis Methods of Cardiac MRI in Assessment of Estimated Corrected Ejection Fraction in Valvular Heart Disease.
Brief Title: Different Methods of Cardiac MRI in Assessment of Estimated Corrected Ejection Fraction in Valvular Heart Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Sous Habib, Resident Doctor, Assiut University
Other Study IDs: Cardiac MRI
Record Dates: First submitted 2023-03-30; First posted 2023-04-11 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Valvular Heart Disease Stenosis and Regurgitation
Keywords: Cardiac MRI methods
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparative study between Phase Contrast , Modified Simpson Rule and Myocardial Strain Analysis methods of Cardiac Magnetic Resonance Imaging in assessment of Corrected Estimated Ejection Fraction in Valvular Heart Disease To Evaluate the diagnostic accuracy of different methods of cardiac MRI to assess estimated corrected ejection fraction in valvular heart diseases.

DETAILED DESCRIPTION:
Valvular heart diseases are common cardiovascular conditions that account for 10% to 20% of all cardiac surgical procedures.

In routine clinical practice,left ventricular performance is one of the most important prognostic factors in valvular heart diseases,whether treated medically or surgically.It gives valuable information that may be useful in the selection of therapy or determination of the optimal time for intervention.

Cardiovascular MR has grown to be a widely used clinical tool for evaluating cardiovascular disease,it is designed to assess cardiovascular morphology,ventricular function,myocardial perfusion,tissue characterization,flow quantification and coronary artery disease.Utilization of CMR for evaluation of valvular regurgitation has recently been recognized as part of the American Society of Echocardiography (ASE) and the Society of Cardiovascular Magnetic Resonance (SCMR) recommendations. In previous guidelines,CMR was only advocated in valvular disease in situations where echocardiographic evaluation was insufficient or inconclusive.However,with excellent spatial and temporal resolution,CMR may provide added benefits for valvular evaluation,including visualization of valve structure, direct measurements of flow,assessment of ventricular volumes, and quantification of regurgitant volumes and fractions .Among CMR techniques are:

* Phase-contrast MRI a technique with which flow can be measured accurately with flexible spatial and temporal resolution .The severity of valvular disease can be assessed and quantified with Phase contrast MRI providing the ability to quantify peak velocities and flow across the valves.
* Simpson rule a method to calculate cardiac global function parameters out of multiple single slices,quantifying volumetric indices of the heart directly from the 3 dimensional dataset; an ability that sets it apart from other modalities. End-Diastolic Volume,End-Systolic Volume,Stroke Volume,Ejection Fraction and Ventricular Mass can be obtained using Simpson rule making it able to determine these measurements in the right side as well as the left.
* Myocardial Strain Analysis provides higher spatial resolution than echocardiography and is useful for the quantitative assessment of cardiac function.Measurement of left ventricular volume parameters such as ejection fraction, end diastolic volume, end systolic volume, stroke volume , cardiac output ,cardiac index and contractile function are possible in analysis using MRI.

ELIGIBILITY:
Inclusion Criteria:

* -All patients referred to radiology departement presented clinically with valvular heart disease.

Exclusion Criteria:

* 1- extremely obese patients. 2-patients with significant issues of claustrophobia. 3- patients with non-MR compatible implants. 4-patients with bad renal function.

Ages: 2 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Normally distributed data will be expressed in form of mean +/- SD and analysed by parametric tests while not normally will be expressed in form of median and analysed by non-parametric tests.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate diagnostic accuracy of different methods of Cardiac MRI to assess valvular heart disease | 2 years 2024-2026
  Cardiac MRI as a diagnostic tool in valvular heart diseases

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A Zaid, Principal Investigator — Assiut University; Ahmed M Hakam, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uretsky S, Wolff SD. Cardiovascular Magnetic Resonance in Valvular Heart Disease-Related Heart Failure. Heart Fail Clin. 2021 Jan;17(1):103-108. doi: 10.1016/j.hfc.2020.09.002. PMID 33220879
- [Background] Blanken CPS, Farag ES, Boekholdt SM, Leiner T, Kluin J, Nederveen AJ, van Ooij P, Planken RN. Advanced cardiac MRI techniques for evaluation of left-sided valvular heart disease. J Magn Reson Imaging. 2018 Aug;48(2):318-329. doi: 10.1002/jmri.26204. PMID 30134000